CLINICAL TRIAL: NCT06514326
Title: The Impact of Mechanisms of Action on Adherence and Outcomes in Unguided Digital Mental Health Interventions: A Randomized Controlled Trial
Brief Title: The Impact of Mechanisms of Action in Unguided Digital Mental Health Interventions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Amit Baumel, Associate Professor, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 418/23
Record Dates: First submitted 2024-07-11; First posted 2024-07-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: DPT-STD; DPT-TP

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPT-STD (Active Comparator): This is the standard intervention arm
  Interventions: Behavioral: DPT-STD
- DPT-TP (Experimental): This is the enhanced intervention arm
  Interventions: Behavioral: DPT-TP

INTERVENTIONS:
Behavioral: DPT-TP — This intervention includes all the ingredients of DPT-STD, but with additional features that correspond to the conceptual model of therapeutic persuasiveness. Each theme in the program comprises a learning phase followed by a 1-2 week focusing phase.
  Accordingly, the program utilizes the following features:
  1. Call to action: Parents receive timely triggers via text messages that are related to the specific goals and therapeutic activities of the modules they have completed.
  2. Monitoring and ongoing feedback of user state: Specific practices currently taught are documented within the system through a brief daily report, on which parents receive feedback.
  3. Adaptation to user state: Parents' reports on their activities are used to acknowledge their success and to suggest additional actions based on the specific goals reported by parents. Effort related to desired therapeutic activities is adapted based on graded tasks.
  Arms: DPT-TP
Behavioral: DPT-STD — This intervention is similar in its features to other programs that deliver DPT, and is suitable for use on computers or on mobile devices. An icon is positioned on the mobile device home screen in order to enable quick access to the program. The DPT-STD comprises seven 10- to 25-minute modules, each corresponding to one of the themes mentioned above. Each module's content includes videos and texts guiding the parent through the training process, and interactive features, such as multiple-choice questions with direct feedback. Additional features embedded within the platform include downloadable materials and a "questions and answers" section that contains frequently asked questions.
  Arms: DPT-STD

SUMMARY:
This randomized controlled trial (RCT) will compare two interventions that utilize the same evidence-based components of established digital parent training programs (DPTs) aimed at treating child behavior problems, but that differ in terms of the quality of therapeutic persuasiveness (TP) quality (standard: DPT-STD; enhanced TP: DPT-TP). The investigators will recruit parents from 160 families with 3-7-year-old children with behavior problems who will be randomized into one of the two intervention arms. The investigators will measure child behavior problems and related parenting variables before, during, and after the intervention. DPT usage will be passively collected.

The investigators hypothesize that, compared to DPT-STD, parents allocated to the DPT-TP arm will have significantly better module completion rates (adherence to the program) and report better outcomes - measured by improvements in child behavior problems and related parenting variables. The investigators also hypothesize that changes in reported outcomes will be mediated by module completion rates. Therefore, comparing two active interventions that only differ in terms of their TP quality will enable to examine the causal link between this conceptual mechanism of action and beneficial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Parents having a child between the ages of 3 and 7
* The parents report high levels of behavior problems demonstrated by their child based on the ECBI Intensity subscale (X ≥ 132)
* The parents have access to a smartphone device with an Internet connection.

Exclusion Criteria:

* The child is taking medication for behavioral or emotional problems
* The child is in regular contact with a professional for behavioral or emotional problems
* their child has been diagnosed with an intellectual disability or developmental delay
* The parents are currently accessing parenting support elsewhere

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Eyberg Child Behavior Inventory (ECBI) | From baseline to 6 months follow-up
  Child behavior problems will be assessed using the Intensity subscale of the 36-item ECBI. For each item, caregivers rate the intensity of the behavior (1 = never to 7 = always).

SECONDARY OUTCOMES:
The Parenting Scale (PS) | From baseline to 6 months follow-up
  Parental disciplinary behaviors in response to their child's misbehaviors will be assessed using two PS subscale scores, Over-reactivity (11 items) and Laxness (10 items), which reflect effective discipline and discipline mistakes on either end, using a 7-point Likert scale.
Alabama Parenting Questionnaire (APQ) | From baseline to 6 months follow-up
  One dimension of parenting practices will be assessed using the APQ Positive Parenting Practices subscale (6 items). Parents will be asked to rate each item on a scale of 1 (never) to 5 (always) according to how often it typically occurs in their home.
The Parenting Tasks Checklist (PTC) | From baseline to 6 months follow-up
  Task-specific self-efficacy will be assessed using 6 items taken from the Behavioural Self-Efficacy PTC subscale. Item responses are given on a scale of 0 (Certain I can't do it) to 100 (Certain I can do it).
Parental Self Efficacy (Me as a Parent [MaaP]) | From baseline to 6 months follow-up
  Overall self-efficacy will be assessed using the 4-item Self-Efficacy subscale of MaaP. Sample items include "I have confidence in myself as a parent" and "My parenting skills are effective." Each item is rated on a Likert scale (1 = strongly disagree; 5 = strongly agree).
Specific Parenting Practices (SPP) | From baseline to 6 months follow-up
  Specific Parenting Practices will be assessed using 12 items that ask about the skills parents acquire directly during the intervention. For example, a sample item targeting the practice of 'recognizing positive behaviors in your child' asks: 'To what extent were you able to express open appreciation and reinforce your child for a specific positive behavior demonstrated?' Parents will be asked to rate how often they demonstrated the expected skill in the past two weeks on a Likert scale (1 = Never; 7 = Always).
Behavior and Feelings Survey (BFS) | From baseline to 6 months follow-up
  The BFS-Internalizing Problems Caregiver version will be used to capture parents report on their childs emotional problems (e.g. anxiety and sadness). It is based on 6 items that are rated on a scale from 0 (not a problem) to 4 (a very big problem).
Program Completion | From baseline to 10 weeks time
  Program completion will be measured based on the percentage of learning modules completed by parents within their respected intervention Arm.

OTHER OUTCOMES:
Minutes of use-Program usage | From baseline to 10 weeks time
  Minutes of use refers to the number of minutes users were logged into the program
Number of logins-Program usage | From baseline to 10 weeks time
  number of unique logins refers to the number of times the user logged into the program
Unique days-Program usage | From baseline to 10 weeks time
  The number of unique days in which the user logged in will be counted
Phases completed | From baseline to 10 weeks time
  The exact learning modules completed by the parents will be documented

CONTACTS AND LOCATIONS:
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baumel A, Aderka IM. The Impact of Mechanisms of Action on Adherence and Outcomes in Self-Guided Digital Mental Health Interventions: Protocol for a Randomized Controlled Trial With Mediation Analysis. JMIR Res Protoc. 2025 May 21;14:e71238. doi: 10.2196/71238. PMID 40397492